CLINICAL TRIAL: NCT03952962
Title: Tractography Guided Subcallosal Cingulate Deep Brain Stimulation for Treatment Resistant Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nader Pouratian (Other)
Responsible Party: Sponsor-Investigator, Nader Pouratian, PROFESSOR & CHAIR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 19-000767; STU-2021-0635
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Treatment Resistant Depression; Undergoing Deep Brain Stimulation (DBS) Surgery
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Intervention Model Description: There will be an initial 12-month open label period for all participants involved. In the second period of the study, patients will be divided into groups: responders (defined as a 40% reduction or more in MADRS) versus non-responders. Responders will continue to the 6-month double-blinded discontinuation phase (see below for additional details of study procedures during this phase). The non-responders, after the open label period (12 months) will have monthly follow-up visits for 12 mo. During the discontinuation period, patients will be randomized to either the ON or OFF stimulation phase for 3 mo each. If randomized to ON, there will be no change for 3 mo, then a biweekly 25% reduction in stimulation amplitude for the next 3 mo until stimulation is off. If randomization to OFF phase, there will be an initial biweekly 25% reduction in stimulation amplitude for 3 mo until the device is off then the stimulation settings will be turned back to the optimized settings for three months.
Masking Description: The investigators propose a clinical trial involving 12-months open-label bilateral DBS that targets SCC (using TOT) in subjects with TRD. The open label period is intended to ensure that maximal benefit can be achieved with the current proposed protocol.
  Following open label optimization, to control for possible placebo, each subject will enter a double blinded randomized discontinuation, intended to confirm clinical benefit of DBS among responders (6 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Randomized Discontinuation Period: OFF then ON DBS (Experimental): Subjects randomized to this arm are initially "OFF" DBS after the open label period then gradually decreased in their optimized setting's amplitude for 8 weeks and then "ON" DBS for 8 weeks.
  Interventions: Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system
- Randomized Discontinuation Period: ON then OFF DBS (Experimental): Subjects randomized to this arm are initially "ON" DBS with optimized stimulation settings for 8 weeks after the open label period and then "OFF" DBS with gradually decreasing amplitude for 8 weeks.
  Interventions: Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system

INTERVENTIONS:
Device: Abbott Laboratories Infinity™ implantable deep brain stimulation system — Deep brain stimulation (DBS) refers to the process of delivering an electrical current to a precise location in the brain.

SUMMARY:
Treatment resistant depression remains a major problem for individuals and society. Surgical procedures may provide relief for some of these patients. The most frequently considered surgical approach is deep brain stimulation (DBS) of a part of the brain called the subcallosal cingulate region. However, the effectiveness and safety is not well established. The investigators will use a novel approach using advanced imaging technique (magnetic resonance tractography) to evaluate the feasibility and safety of this surgical approach. An innovative method for the definition of DBS target will be applied that redefines the concept of targeting as one of targeting a symptomatic network rather than a structural brain region using subject-based brain anatomy to define the target location. The correlation between imaging findings at baseline with the mood score changes at different time points of the study will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (non-pregnant) between ages 21 and 70;
* DSM-5 diagnosis a current major depressive episode (MDE) for 10 years of less, recurrent or single episode with first episode after adulthood and did not start during childhood or adolescence, secondary to nonpsychotic unipolar major depressive disorder;
* Current index MDE ≥24 months duration and/or recurrent illness with at least a total of 2 lifetime episodes (including current episode >12 months);
* Treatment resistance (defined by criteria on the Antidepressant Treatment History Form (ATHF)28): Failure to respond to a minimum of four adequate depression treatments from different categories;
* Symptom severity for Screening: Hamilton Depression Rating Scale-17 item (HDRS17) ≥20;
* Symptom severity for Outcome: Montgomery Asberg Rating Scale (MADRS) ≥27 to be met at assessment one week pre-op;
* Normal brain MRI within 3 months of surgery;
* Antidepressant medication regimen has been held stable for ≥ 30 days prior to the study screening MADRS;
* Remain on stable antidepressant medication throughout the study, unless there are safety concerns;
* Montreal Cognitive Assessment (MoCA) >25;
* Able and willing to give informed consent and agree to attend regular clinic visits for at least 12 months.

Exclusion Criteria:

* DSM-5 Axis I Disorders: any lifetime history of psychotic disorder or bipolar disorder;
* Alcohol or substance use disorder within 6 months, excluding nicotine;
* History of childhood abuse (physical or sexual) 18
* Personality disorders;
* Seeking disability during the trial;
* Current substantial suicidal risk as defined by a plan or clear immediate intent for self-harm, or made any suicide attempt within the last year; (MADRS ≥ 5 including the day of surgery);
* No stable work history;
* Neurological/Medical condition that makes the patient, in the opinion of the surgeon, a poor candidate;

  1. Pregnant or has plans to become pregnant in the next 36 months;
  2. Unable/unable to practice birth control through the period of randomization and withdrawal of therapy;
* Subjects who have a history of a seizure disorder;
* Subjects who will be exposed to diathermy;
* Subjects who have any medical contraindications to undergoing DBS surgery (e.g. infection, coagulopathy, or significant cardiac or other medical risk factors for surgery);
* Subjects with another implanted device such as a cardiac pacemaker, defibrillator or neurostimulator;
* Subjects who have a history of hemorrhagic stroke;
* Subjects who are unable to undergo MRI;
* Subjects who are at increased risk of hemorrhage due to underlying medical conditions or medication.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery and Asberg Depression Rating Scale (MADRS) score. | 18 months
  The primary endpoint will be defined as at least a 40% reduction in the Montgomery and Asberg Depression Rating Scale (MADRS) that measures depression severity. The MADRS scores range from 0 to 60, where increased values indicate more severe depression. There are 10 questions that each yield a score of 0-6 that are then summed for a total score.

SECONDARY OUTCOMES:
Change in another related clinical assessment: PHQ-9 | 18 months
  Change in PHQ-9: Patient Health Questionnaire 9. The PHQ-9 the 9-item depression module from the full PHQ. Major depression is diagnosed if 5 or more of the 9 depressive symptom criteria have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. Other depression is diagnosed if 2, 3, or 4 depressive symptoms have been present at least "more than half the days" in the past 2 weeks, and 1 of the symptoms is depressed mood or anhedonia. One of the 9 symptom criteria ("thoughts that you would be better off dead or of hurting yourself in some way") counts if present at all, regardless of duration. The clinician is expected to rule out physical causes of depression, normal bereavement, and history of a manic episode. As a severity measure, the PHQ-9 score can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Change in another related clinical assessment: QIDS-SR | 18 months
  Change in QIDS-SR: Quick Inventory of Depressive Symptomatology Self Report. The QIDS-SR is a 16-question shortened self-test, derived from the 30-item Inventory of Depressive Symptomatology (IDS), which measures 9 different criterion domains of major depression. Each of the 4 possible answers to each quiz is given an ascending numerical value from 0-3, where increased values indicate the severity of depressive symptom.
Change in another related clinical assessment: HAM-A | 18 months
  Change in HAM-A: Hamilton Anxiety Rating Scale. The HAM-A is a 14-item test designed to assess the severity of anxiety symptoms. All questions are rated on a 5-point (0-4) scale, with 7 questions on psychic anxiety and 7 questions on somatic anxiety. Total scores range from 0 to 56. Patients with anxiety and panic disorder tend to have a score greater than 20.
Change in another related clinical assessment: CSSRS | 18 months
  Change in CSSRS: Columbia Suicide-Severity Rating Scale. The C-SSRS is a semistructured clinical interview that utilizes a set of prompts and questions to help an interviewer get more complete information on events suggestive of suicidality. This prospective tool aims to standardize terminology and articulate suicidality assessment in a straightforward manner. The categories within the assessment involve binary responses (yes/no) that establish the intensity of suicide ideation on a scale of 1-5, where 5 is most severe.
Change in another related clinical assessment: HAMD-17 | 18 months
  Change in HAMD-17:Hamilton Rating Scale for Depression. The HAMD-17 is a 17-item scale that evaluates depressed mood, vegetative and cognitive symptoms of depression, and comorbid anxiety symptoms. The HAMD-17 was one of the first rating scales developed to quantify the severity of depressive symptomatology. First introduced by Max Hamilton in 1960, it has since become the most widely used and accepted outcome measure for evaluating depression severity. It provides ratings on current DSM-IV symptoms of depression, with the exceptions of hypersomnia, increased appetite, and concentration/indecision. The HAMD-17 was designed to be administered by a trained clinician using a semi-structured clinical interview. The 17- items are rated on either a 5-point (0-4) or a 3-point (0-2) scale.
Change in another related clinical assessment: SCID-II | 18 months
  Change in SCID-II: Structural Clinical Interview for Personality Disorders.This is a semi-structured interview for making DSM-IV Axis II (Personality Disorder) diagnoses and is designed to be administered by a clinician or trained mental health professional. A SCID II takes 1/2 to 1 hour to administer. There are 3 components to the SCID-II. The interview itself covers the 11 DSM-IV Personality Disorders. After the subject fills out the Personality Questionnaire (which usually takes 20 minutes), the clinician simply circles the numbers to the left of the SCID-II items that correspond to items answered "yes" on the questionnaire. The clinician needs only to inquire about the items screened positive on the questionnaire. The assumption is that a subject who responds with a "no" on the questionnaire item would also have answered "no" to the same question had it been read aloud by the interviewer. For this study, only the subsection for Cluster B will be administered.
Change in another related clinical assessment: CGI | 18 months
  Change in CGI: Clinical Global Impression of Severity and Improvement. The CGI is used to measure the global impression of a treatment response in a psychiatric patient's illness by a clinician. Two of three sub-scales are being used to measure severity of the illness and improvement of the illness. Items in the two-subscales being administered are rated on a seven-point scale ranging from "1=normal" to "7=extremely ill" for severity subscale and "1=very much improved" to "7=very much worse" for improvement sub-scale.
Change in another related clinical assessment: PGI | 18 months
  Change in PGI: Patient Global Impression Index. The PGI is used to measure the global impression of a treatment response in a psychiatric patient's illness by the patient. Two sub-scales are being used to measure severity of the illness and improvement of the illness. Items in the two-subscales being administered are rated on a seven-point scale ranging from "1=normal not ill at all" to "7=among the most extremely ill" for severity sub-scale and "1=very much improved" to "7=very much worse" for improvement sub-scale.
Change in another related clinical assessment: MoCA | 18 months
  Change in MoCA: Montreal Cognitive Assessment. The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Change in another related clinical assessment: SAFTEE-SI | 18 months
  Change in SAFTEE-SI: Systematic Assessment for Treatment Emergent Events - Specific . The SAFTEE is a structural clinical interview developed by the National Institute of Mental Health which exams possible treatment-emergent side effects for clinical studies. The SAFTEE-SI looks at specific adverse symptoms for a particular treatment/ clinical trial where the summary scores represent the number of adverse events experienced.
Change in another related clinical assessment: SF-36 | 18 months
  Change in SF-36: Short Form 36. The SF-36 Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status and is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change in another related clinical assessment: QOL | 18 months
  Change in QOL: Quality of Life Enjoyment and Satisfaction Questionnaire. The short form of the QOL is a self-report form composed of 16 items each rated on a 5-point scale that indicates the degree of enjoyment or satisfaction experienced during the past week. A total score of items 1 to 14 is computed and expressed as a percentage of the maximum possible score of 70. The 14 items evaluated each subjects' satisfaction with his or her physical health, social relations, ability to function in daily life; ability to get around physically; mood; family relations; sexual drive and interest; ability to work on hobbies, work, leisure time activities; economic status; household activities; living/housing situation; and overall sense of well-being.
Change in another related clinical assessment: HLQ | 18 months
  Change in HLQ: Health and Labor Questionnaire. The HLQ is designed to collect quantitative data on the relation between illness and treatment and work performance. The HLQ data permits the estimation of production losses (costs) of paid and unpaid labor. It contains also an indicator for impediments for paid and unpaid labor, one of the indicators for quality of life. The HLQ is divided into 4 modules to collect data about absence from work, reduced productivity at paid work, unpaid labor production and impediments to paid and unpaid labor. The modular structure permits the omission of questions that are not applicable to the study population. The questionnaire is suitable for self-assessment.
Change in another related clinical assessment: YMRS | 18 months
  Change in YMRS: Young Mania Rating Scale. The Young Mania Rating Scale (YMRS) is a rating scale to assess manic symptoms. The scale has 11 items and is based on the patient's subjective report of their clinical condition over the previous 48 hours. The items are selected based upon published descriptions of the core symptoms of mania. Each item given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. The authors encourage the use of whole or half point ratings once experience with the scale is acquired. Typical baseline scores can vary a lot and depend on the patients' clinical features such as mania (YMRS = 12), depression (YMRS = 3), or euthymia (YMRS = 2). Sometimes a clinical study entry requirement of YMRS > 20 generates a mean YMRS baseline of about 30.
Change in another related clinical assessment: PSQI | 18 months
  Change in PSQI: Pittsburgh Sleep Quality Index. The PSQI is a 19-item questionnaire evaluating sleep quality and disturbances over the past month.The first 4 items are open questions, whereas items 5 to 19 are rated on a 4-point Likert scale. Individual items scores yield 7 components. A total score, ranging from 0 to 21, is obtained by adding the 7 component scores. A score > 5 suggests poor sleep quality. The psychometric properties of the PSQI have been documented in multiple studies, including one with a French-Canadian sample. The PSQI was used because it measures a construct (sleep quality) that is related to insomnia but a construct that is broader than insomnia severity. It was administered to the community sample only.
Change in another related clinical assessment: ISI | 18 months
  Change in ISI: Insomnia Severity Index. The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia. The usual recall period is the "last month" and the dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia (22-28). Three versions are available-patient, clinician, and significant others-but the present paper focuses on the patient version only.
Change in another related clinical assessment: LAPS | 18 months
  Change in LAPS: Leuven Affect and Pleasure Scale. The LAPS is a comprehensive depression assessment scale that integrates several theoretical frameworks on negative and positive affect an on anhedonia. The LAPS comprising of 16 items grouped in 6 categories addresses not only negative affects (depressed mood and anxiety) but also the positive affects, anhedonia, cognitive and overall functioning on a scale of 0-10, where 10 is very much experiencing a feeling/ affect and 0 is not at all.
Change in another related clinical assessment: SHAPS | 18 months
  Change in SHAPS: Snaith-Hamilton Pleasure Scale. The 14-item SHAPS is a self-administered instrument that was used to measure hedonic experience or positive valence. Each of the items has a set of four response categories--Strongly Agree, Agree, Disagree, and Strongly Disagree, with either of the Agree responses receiving a score of 0 and either of the Disagree responses receiving a score of 1. Total scores ranged from 0 to 14, with higher scores indicating a lower level of hedonic experience or a higher level of anhedonia.
Change in another related clinical assessment: TEPS | 18 months
  Change in TEPS: Temporal Experience of Pleasure Scale. The TEPS has 18 items and two subscales designed to distinguish between anticipatory and consummatory pleasure. It uses a 6-point Likert scale (from 1 = very false for me to 6 = very true for me). Items only reflect physical anhedonia. A significant advantage of this scale is that its two-factor structure that separates anticipatory and consummatory aspects of reward.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Pouratian, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Investigators with established research programs will be eligible for data sharing. Interested investigators will be required to submit a summary of proposed work and requested data elements. If approved by the Principal Investigator of the study, data will be shared. This data will be de-identified and coded. There is no plan to share identifiers outside the study team